CLINICAL TRIAL: NCT02998671
Title: A Randomized, Subject and Investigator Blinded, Placebo-controlled, Multi-center Study in Parallel Groups to Assess the Efficacy and Safety of CJM112 in Patients With Moderate to Severe Inflammatory Acne
Brief Title: Study of Efficacy and Safety of CJM112 in Patients With Moderate to Severe Inflammatory Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCJM112X2203
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Acne Vulgaris
Keywords: Acne, inflammatory acne, efficacy, safety, PK
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: CJM112 high dose (Experimental): CJM112 high dose in treatment period 1; CJM112 high dose in extension period 2
  Interventions: Biological: CJM112
- Group 2: CJM112 low dose (Experimental): CJM112 low dose in treatment period 1; CJM112 low dose in extension period 2
  Interventions: Biological: CJM112
- Group 3: Placebo, CJM112 low dose or high dose (Placebo Comparator): Placebo in treatment period 1; CJM112 low dose or CJM112 high dose in extension period 2
  Interventions: Biological: CJM112; Other: Placebo

INTERVENTIONS:
Biological: CJM112
Other: Placebo
  Arms: Group 3: Placebo, CJM112 low dose or high dose

SUMMARY:
The study was designed primarily to assess preliminary efficacy and safety of CJM112 in patients with moderate to severe inflammatory acne and to determine if CJM112 has an adequate clinical profile for further clinical development. In addition, sustainability of response and dose relationship were to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 45 years of age included, and otherwise in good health as determined by medical history, physical examination, vital signs, ECGs and laboratory tests at screening.
* Body weight between 50 and 120 kg, inclusive at screening.
* Patients with papulo-pustular acne vulgaris with between 25 and 100 facial inflammatory lesions (papules, pustules and nodules), and presence of non-inflammatory lesions (open and closed comedones) in the face at screening and baseline, who have failed systemic therapy for inflammatory acne.
* No more than 5 facial inflammatory nodules at screening and baseline.
* Investigator's Global assessment (IGA) score of at least moderate (3) acne severity on the face at screening and baseline.

Exclusion Criteria:

* Appropriate wash out periods are required for investigational drugs, any oral/systemic treatment for acne, systemic or lesional injected (for acne) corticosteroids or systemic immunomodulators, any systemic hormonal treatments, previous treatment with biologics, oral retinoids (in particular isotretinoin) and any topical anti-acne treatment.
* Use of facial medium depth chemical peels (excluding home regimens) within 3 months prior to baseline.
* Any live vaccines (this includes nasal-spray flu vaccine) starting from 6 weeks before baseline.
* Any other forms of acne
* Any severe, progressive or uncontrolled medical or psychiatric condition or other factors at randomization that in the judgment of the investigator prevents the patient from participating in the study.
* History of hypersensitivity or allergy to the investigational compound/compound class being used in this study.
* Active systemic infections (other than common cold) during the 2 weeks prior to baseline.
* History of severe systemic Candida infections or evidence of Candidiasis in the 2 weeks prior to baseline.
* Evidence of active tuberculosis at screening. All patients will be tested for tuberculosis status using a blood test (QuantiFERON®-TB (Tuberculosis) Gold In-Tube). Patients with evidence of tuberculosis may enter the trial afteradequate treatment has been started according to local regulations.
* Patients with known active Crohn's disease
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result at screening.
* A positive Hepatitis B surface antigen or Hepatitis C test result at screening
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human chorionic gonadotropin (HCG) laboratory test.
* WOCBP, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 13 weeks after stopping medication.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Novartis Investigative Site, Culver City, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Austin, Texas
- Germany (4):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Pommelsbrunn
- Netherlands (3):
  - Novartis Investigative Site, Bergen op Zoom
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiden

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of approximately 75 subjects were planned to be enrolled in the study. The study was terminated early due to futility after a total of 52 subjects were enrolled and randomized.
Pre-assignment Details: For period 1 (12 weeks) subjects were randomized to one of the 3 treatment groups CJM112 high dose, CJM112 low dose or placebo.
  For Period 2 (12 weeks) subjects treated with Placebo in Period 1 were rerandomized to CJM112 high dose or CJM112 low dose. All other subjects remained on the same dose.
Groups:
- P1: CJM112 High Dose / P2: CJM112 High Dose: CJM112 high dose (300mg) in treatment period 1 (Day 1 - 85) ; CJM112 high dose (300mg) in extension period 2 (Day 86 - 169)
- P1: CJM112 Low Dose / P2: CJM112 Low Dose: CJM112 low dose (75mg) in treatment period 1 (Day 1 - 85) ; CJM112 low dose (75mg) in extension period 2 (Day 86 - 169)
- P1: Placebo / P2: CJM112 High Dose: Placebo in treatment period 1 (Day 1 - 85); CJM112 high dose (300mg) in extension period 2 (Day 86 - 169)
- P1: Placebo / P2: CJM112 Low Dose: Placebo in treatment period 1 (Day 1 - 85) ; CJM112 low dose (75mg) in extension period 2 (Day 86 - 169)
- P1: Placebo / P2: NA: Placebo in treatment period 1 (Day 1 - 85); Patients did not enter extension period 2
Period: Period 1
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA
Started | 21 | 13 | 6 | 8 | 4
Completed | 17 | 10 | 6 | 8 | 0
Not Completed | 4 | 3 | 0 | 0 | 4
Not completed — Study Terminated By Sponsor | 2 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA
Started | 17 | 10 | 6 | 8 | 0
Completed | 14 | 3 | 5 | 4 | 0
Not Completed | 3 | 7 | 1 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 3 | 5 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA | Total
Number analyzed (Participants) | 21 | 13 | 6 | 8 | 4 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (4.19) | 25.5 (5.99) | 22.5 (3.21) | 25 (4.66) | 23.75 (4.35) | 24.3 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 3 | 6 | 4 | 34
  Male | 8 | 5 | 3 | 2 | 0 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 10 | 5 | 8 | 4 | 45
  Other | 3 | 3 | 1 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Inflammatory Facial Lesion Count at Day 85
Description: Total inflammatory facial lesion count was the total count of papules, pustules and nodules assessed at day 85
Time Frame: Day 85
Population: Pharmacodynamic analysis set, including only patients completing 12-week assessments.
Measure: Geometric Mean (90% Confidence Interval); unit: Lesions
Groups:
- P1: Placebo / P2 CJM112 Low Dose or High Dose: Placebo in treatment period 1 (Day 1 - 85) ; CJM112 low dose or CJM112 high dose in extension period 2 (Day 86 - 169)
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2 CJM112 Low Dose or High Dose
Number analyzed (Participants) | 17 | 10 | 15
Lesions | 21.9 [16.58 to 29.14] | 20.3 [13.76 to 29.66] | 18.5 [13.51 to 25.13]
Statistical Analysis 1: Comparison: P1: CJM112 High Dose / P2: CJM112 High Dose vs P1: Placebo / P2 CJM112 Low Dose or High Dose; Test type: Superiority — Comparison at end of Period 1 (P1): CJM112 versus Placebo; Bayesian model for repeated measurements; Ratio of geometric means = 1.18, 90% CI 2-sided [0.79 to 1.81] — Ratio of Geometric Means (CJM112 / Placebo) calculated. A value > 1 indicates a higher number of lesion counts in the CJM112 group. Bayesian analysis. The "credible interval" was calculated and presented under "confidence interval"
Statistical Analysis 2: Comparison: P1: CJM112 Low Dose / P2: CJM112 Low Dose vs P1: Placebo / P2 CJM112 Low Dose or High Dose; Test type: Superiority — Comparison at end of Period 1 (P1): CJM112 versus Placebo; Bayesian model for repeated measurements; Ratio of geometric means = 1.10, 90% CI 2-sided [0.66 to 1.80] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number and Severity of Adverse Events in Period 1
Description: Frequency and severity of adverse events in Period 1
Time Frame: Day 1 to Day 85
Population: Safety analysis set
Measure: Number; unit: Adverse Events
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2 CJM112 Low Dose or High Dose
Number analyzed (Participants) | 21 | 13 | 18
Adverse Events
  Number of AEs of mild intensity | 27 | 25 | 20
  Number of AEs of moderate intensity | 5 | 7 | 9
  Number of AEs of severe intensity | 0 | 1 | 0

3. Secondary Outcome: Number and Severity of Adverse Events in Period 2
Description: Frequency and severity of adverse events in Period 2
Time Frame: Day 86 to Day 260
Population: Safety analysis set
Measure: Number; unit: Adverse Events
Groups:
- P1: Placebo / P2: CJM112 High Dose: Placebo in treatment period 1; CJM112 high dose in extension period 2
- P1: Placebo / P2: CJM112 Low Dose: Placebo in treatment period 1; CJM112 low dose in extension period 2
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose
Number analyzed (Participants) | 17 | 10 | 6 | 8
Adverse Events
  Number of AEs of mild intensity | 21 | 20 | 6 | 13
  Number of AEs of moderate intensity | 6 | 1 | 3 | 1
  Number of AEs of severe intensity | 1 | 1 | 0 | 0

4. Secondary Outcome: Pharmacokinetics (PK): Serum Trough Concentrations of CJM112 in Period 1
Description: Pharmacokinetics (PK): Serum trough concentrations of CJM112. Concentrations below the lower limit of quantification were reported as 0.
Time Frame: Day 1, Day 29, Day 57 and Day 85
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose
Number analyzed (Participants) | 21 | 12
ng/mL
  Period 1 Day 1 (Pre Dose): number analyzed (Participants) | 19 | 11
  Period 1 Day 1 (Pre Dose) | 152 (663) | 0 (0)
  Period 1 Day 29 (Pre Dose): number analyzed (Participants) | 20 | 11
  Period 1 Day 29 (Pre Dose) | 8670 (3370) | 802 (961)
  Period 1 Day 57 (Pre Dose): number analyzed (Participants) | 19 | 10
  Period 1 Day 57 (Pre Dose) | 11500 (5020) | 1550 (1130)
  Period 1 Day 85 (Pre Dose): number analyzed (Participants) | 16 | 9
  Period 1 Day 85 (Pre Dose) | 17000 (8080) | 2040 (1570)

5. Secondary Outcome: Pharmacokinetics (PK): Serum Trough Concentrations of CJM112 in Period 2
Description: as for outcome 4
Time Frame: Day 85, Day 113, Day 141 and Day 169
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose
Number analyzed (Participants) | 21 | 12 | 6 | 8
ng/mL
  Period 2 Day 85 (Pre Dose): number analyzed (Participants) | 16 | 9 | 6 | 8
  Period 2 Day 85 (Pre Dose) | 17000 (8080) | 2040 (1570) | 713 (1750) | 0 (0)
  Period 2 Day 113 (Pre Dose): number analyzed (Participants) | 16 | 6 | 6 | 7
  Period 2 Day 113 (Pre Dose) | 15900 (8140) | 1890 (634) | 8260 (5120) | 1430 (1190)
  Period 2 Day 141 (Pre Dose): number analyzed (Participants) | 16 | 3 | 5 | 6
  Period 2 Day 141 (Pre Dose) | 18700 (9450) | 3140 (2180) | 15700 (10700) | 3700 (1250)
  Period 2 Day 169 (Pre Dose): number analyzed (Participants) | 14 | 3 | 5 | 4
  Period 2 Day 169 (Pre Dose) | 19400 (9650) | 3890 (1890) | 16600 (6610) | 2890 (672)

6. Secondary Outcome: Number of Patients With Clinically Significant Abnormal Hematology Laboratory Parameters
Description: Abnormalities were considered clinically significant by the Investigator if they could impact the study conduct or safety of the subjects.
Time Frame: 38 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA
Number analyzed (Participants) | 21 | 13 | 6 | 8 | 4
Participants
  Period 1 | 0 | 0 | 0 | 0 | 0
  Period 2: number analyzed (Participants) | 17 | 10 | 6 | 8 | 0
  Period 2 | 0 | 0 | 0 | 0 |

7. Secondary Outcome: Number of Patients With Clinically Significant Abnormal Clinical Chemistry Laboratory Parameters Parameters
Description: as for outcome 6
Time Frame: 38 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA
Number analyzed (Participants) | 21 | 13 | 6 | 8 | 4
Participants
  Period 1 | 3 | 0 | 0 | 0 | 0
  Period 2: number analyzed (Participants) | 17 | 10 | 6 | 8 | 0
  Period 2 | 0 | 3 | 1 | 1 |

8. Secondary Outcome: Number of Patients With Clinically Significant Abnormal Urinalysis Laboratory Parameters
Description: as for outcome 6
Time Frame: 38 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | P1: CJM112 High Dose / P2: CJM112 High Dose | P1: CJM112 Low Dose / P2: CJM112 Low Dose | P1: Placebo / P2: CJM112 High Dose | P1: Placebo / P2: CJM112 Low Dose | P1: Placebo / P2: NA
Number analyzed (Participants) | 21 | 13 | 6 | 8 | 4
Participants
  Period 1 | 0 | 0 | 0 | 0 | 0
  Period 2: number analyzed (Participants) | 17 | 10 | 6 | 8 | 0
  Period 2 | 0 | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: 38 weeks
Groups:
- Period 1: CJM112 High Dose: Period 1: CJM112 high dose (300mg)
- Period 1: CJM112 Low Dose: Period 1: CJM112 low dose (75mg)
- Period 1: Placebo: Period 1: Placebo
- Period 1: Pooled CJM112: Period 1: Pooled CJM112
- Period 2: CJM112 High Dose/CJM112 High Dose: CJM112 high dose (300mg) in treatment period 1; CJM112 high dose (300mg) in extension period 2
- Period 2: CJM112 Low Dose/CJM112 Low Dose: CJM112 low dose (75mg) in treatment period 1 ; CJM112 low dose (75mg) in extension period 2
- Period 2: Placebo/ CJM112 High Dose: Placebo in treatment period 1; CJM112 high dose (300mg) in extension period 2
- Period 2: Placebo/ CJM112 Low Dose: Placebo in treatment period 1; CJM112 low dose (75mg) in extension period 2
- Period 2: Pooled CJM112 High Dose: Period 2: Pooled CJM112 high dose (300mg)
- Period 2: Pooled CJM112 Low Dose: Period 2: Pooled CJM112 low dose (75mg)
Arm/Group | Period 1: CJM112 High Dose | Period 1: CJM112 Low Dose | Period 1: Placebo | Period 1: Pooled CJM112 | Period 2: CJM112 High Dose/CJM112 High Dose | Period 2: CJM112 Low Dose/CJM112 Low Dose | Period 2: Placebo/ CJM112 High Dose | Period 2: Placebo/ CJM112 Low Dose | Period 2: Pooled CJM112 High Dose | Period 2: Pooled CJM112 Low Dose
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/13 | 0/18 | 0/34 | 0/17 | 0/10 | 0/6 | 0/8 | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/13 | 0/18 | 0/34 | 1/17 | 0/10 | 0/6 | 0/8 | 1/23 | 0/18
Other Adverse Events (participants affected / at risk) | 16/21 | 11/13 | 10/18 | 27/34 | 10/17 | 9/10 | 5/6 | 5/8 | 15/23 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: CJM112 High Dose (N=21) | Period 1: CJM112 Low Dose (N=13) | Period 1: Placebo (N=18) | Period 1: Pooled CJM112 (N=34) | Period 2: CJM112 High Dose/CJM112 High Dose (N=17) | Period 2: CJM112 Low Dose/CJM112 Low Dose (N=10) | Period 2: Placebo/ CJM112 High Dose (N=6) | Period 2: Placebo/ CJM112 Low Dose (N=8) | Period 2: Pooled CJM112 High Dose (N=23) | Period 2: Pooled CJM112 Low Dose (N=18)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: CJM112 High Dose (N=21) | Period 1: CJM112 Low Dose (N=13) | Period 1: Placebo (N=18) | Period 1: Pooled CJM112 (N=34) | Period 2: CJM112 High Dose/CJM112 High Dose (N=17) | Period 2: CJM112 Low Dose/CJM112 Low Dose (N=10) | Period 2: Placebo/ CJM112 High Dose (N=6) | Period 2: Placebo/ CJM112 Low Dose (N=8) | Period 2: Pooled CJM112 High Dose (N=23) | Period 2: Pooled CJM112 Low Dose (N=18)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 4 | 2 | 1 | 0 | 2 | 2 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02998671/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02998671/SAP_001.pdf